CLINICAL TRIAL: NCT03848975
Title: Impact of Simulation Training on the Success Rate of External Cephalic Version and Vacuum Assisted Delivery in Clinical Practice. A Randomized Controlled Trial.
Brief Title: Impact of Simulation Training for Obstetrics-gynecology Residents.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Nicole Jastrow Meyer, Principal investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-00310
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Simulation Training
Keywords: Simulation training; Obstetrics; External cephalic version; Vacuum assisted delivery

STUDY DESIGN:
Intervention Model Description: For the intervention (trained) group, training sessions will be conducted over six months. The control group will learn obstetric maneuver during daily clinical practice in the delivery room under supervision (usual resident training without simulation sessions). The groups will "cross-over" for the next 6 months.
  After six months the success rate and secondary outcomes will be analyzed. The comparison will be, first, between the intervention (trained) group and the control group and, second, for each subject, between its success rate reported before and its success rate after the observation period.
  Some aspects of our study design can be those of a cross over trial, or a stepped wedge design : the participants will have intervention ECV followed, after 6 months, by intervention VE, or intervention VE followed, after 6 months, by intervention ECV. However as some aspects are not those of the above designs, the investigators believe that the best category is a parallel trial.
Masking Description: The person who generate the randomization list and prepare the envelopes will not be involved later in the study. The subject of this study necessarily involves the fact that the participants know the group to which they are assigned. They will be asked to avoid to reveal their allocation to the other care providers (midwives and other colleagues) involved in the care of the patients delivering under their supervision. The investigator responsible for collecting and coding the data will not know to which group belongs the person being evaluated. In some cases, the midwife in charge of the patient will collect the data. She will not know to which group belongs to the person being evaluated. The patient will not know to which group belongs the doctor practicing the obstetric maneuver. However the study taking place within a hospital, it can not be excluded that a care provider or an outcome assessor learns informally the allocation of one or more participants, despite these precautions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulation training for ECV (Experimental): For the intervention (trained) group, the training sessions will be conducted over six months. During this period participants will continue their daily clinical practice in the delivery room: when one of these maneuvers is needed, a case report form (CRF) will be completed by the participant. This group is the Control group for VE : The control group will learn obstetric maneuver during daily clinical practice in the delivery room under supervision (usual resident training without simulation sessions). When one of these maneuvers is needed, a case report form (CRF) will be completed by the participant.
  Interventions: Other: Simulation training for ECV
- Simulation training for VE (Experimental): For the intervention (trained) group, the training sessions will be conducted over six months. During this period participants will continue their daily clinical practice in the delivery room: when one of these maneuvers is needed, a case report form (CRF) will be completed by the participant. This group is the the control group for for ECV : The control group will learn obstetric maneuver during daily clinical practice in the delivery room under supervision (usual resident training without simulation sessions). When one of these maneuvers is needed, a case report form (CRF) will be completed by the participant.
  Interventions: Other: Simulation training for VE

INTERVENTIONS:
Other: Simulation training for ECV — Intervention for the ECV group is a ECV simulation training. The group will have theoretical courses and five simulation sessions with four ECV simulation on a model (i.e., a total of 20 ECV), associated with clinical practice in the delivery room.
  Arms: Simulation training for ECV
Other: Simulation training for VE — Intervention for the VE group is a simulation training. The group will have theoretical courses and five simulation sessions with four VE simulation on a model (i.e., a total of 20 VE), associated with clinical practice in the delivery room. The investigators will us Kiwi® Omni Cup Vacuum Delivery System, as this is the vacuum system chosen for clinical practice in our obstetric service.
  Arms: Simulation training for VE

SUMMARY:
The main objective of the study is to evaluate the benefit of simulator training for learning external cephalic version (ECV) or vacuum assisted vaginal delivery (hereafter vacuum extraction [VE]) for obstetrics-gynecology residents.

The primary outcome of this randomized control trial is to evaluate the impact of simulation training on the success of ECV and VE.

DETAILED DESCRIPTION:
Usually, the training of obstetrical maneuvers are done "one the job" according to the situations encountered in the clinical practice during postgraduate training. This has some disadvantages like inequality of exposure to these situations, inadequate learning environment (emergencies, impossibility to repeat the maneuver, etc.) and risk complications related to the learner'slack of experience. To evaluate the benefit for learning external cephalic version (ECV) or vacuum assisted vaginal delivery (hereafter vacuum extraction [VE]), the investigators are conducting a randomized control trial composed by two parallel studies. Each group will represent the control group in relation to the maneuver to which it will not be trained.

The objectives of the first one is to evaluate the impact of simulation training on the success of ECV, the complication rate, as well as the patient's and learner's satisfaction. The objectives of the second one is to evaluate the impact of simulation training on the success of VE, the complication rate, as well as the patient's and learner's satisfaction.

The overall goal is to evaluate the effects on clinically relevant outcomes of the teaching by simulation in obstetrics. If simulation training improves the success rate of these maneuvers and the satisfaction of the patient and the learner, simulation learning will be included in a formal and systematic way during postgraduate training in obstetrics.

The subjects are the resident doctors or consultants who have had no or few prior simulation training (maximum 1 session) and little clinical experience of the maneuver evaluated (maximum of 19 of each maneuver).

ELIGIBILITY:
Inclusion Criteria:

* Being a resident or consultant working in the gynecology and obstetrics department of the hospital
* Agreeing to participate in the study by signing an informed consent form

Exclusion Criteria:

* Having performed several ECV or VE simulation training (more than 1 session each) before the recruitment
* Having already performed more than 20 ECV and more than 20 VE during clinical practice before recruitment.
* Having a planned clinical activity in the delivery room which does not allow to perform at least 1 ECV or 1 VE during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2018-08-28 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of the ECV in the participant clinical practice | 6 months
  The success of the procedure is defined as the passage of the fetus from a breech ou transverse presentation to a cephalic presentation, immediately confirmed by ultrasound, after a maximum of 2 trials. The outcomes for each procedure (success or not) will be judged at the end of the procedure
Success rate of the VE in the participant clinical practice | 6 months
  The success rate of the procedure is defined as birth after vacuum-assisted delivery without release of the Kiwi cup. The cup's release is considered when total and involuntary loss of vacuum occurs, resulting in a loss of contact with the head. If the patient gives birth spontaneously after a vacuum release or if there is a change of instrumentation (following a release or not), it is a failure in the context of this study. The outcomes for each procedure (success or not) will be judge at the end of the procedure

SECONDARY OUTCOMES:
Reason for stopping ECV | 6 months
  That is : success, patient request, transmission to supervisor, maximum number of trials reached
Maximum pain during ECV on numeric rating scale | 6 months
  Maximum pain during the procedure, reported by the women, using a the numeric rating scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain)
Maternal satisfaction after the ECV on numeric rating scale | 6 months
  Global satisfaction reported by the women 2 hours after the ECV using a the numeric rating scale. The scale is composed of 1 (very unsatisfied) to 10 (very satisfied)
Participant satisfaction after the ECV on numeric rating scale | 6 months
  Global satisfaction reported by the participant after the ECV using a the numeric rating scale. The scale is composed of 1 (very unsatisfied) to 10 (very satisfied)
Rate of complication (ECV) | 6 months
  That is : bleeding, suspicious or pathological cardiotocography (see appendix 1), Kleihauer> 1, retro-placental hematoma, reported in the hour following the ECV
Rate of emergency cesarean section (ECV) | 6 months
  Rate of emergency cesarean section performed in case of ECV complication
Reason for stopping VE | 6 months
  That is : success, release, transmission to supervisor
Number of pull for VE | 6 months
  Number of pull on the Kiwi® Omni Cup Vacuum Delivery System necessary for birth
Maternal satisfaction after the VE on numeric rating scale | 6 months
  Global satisfaction reported by the women 2 hours after the VE using a the numeric rating scale. The scale is composed of 1 (very unsatisfied) to 10 (very satisfied)
Participant satisfaction after the VE on numeric rating scale | 6 months
  Global satisfaction reported by the participant after the VE using a the numeric rating scale. The scale is composed of 1 (very unsatisfied) to 10 (very satisfied)
Rate of complication (VE) | 6 months
  That is : subdural hematoma, subgaleal or intracranial hemorrhage, skull fracture, fetal scalp laceration, third- or four-degree perineal tear, vaginal tear)
Rate emergency cesarean section rate (VE) | 6 months
  Rate of emergency cesarean section performed and indication

OTHER OUTCOMES:
Cup position (VE) | 6 months
  The investigators will document with a picture of the newborn's skull the area where the cup was placed to determine if the placement of the cup was correct. The photos will then be reviewed by the investigator and the position will be judged correct or incorrect. The correct positioning rate will be calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Gynecology & obstetrics department of Geneva University Hospital (Hôpitaux Universitaires de Genève (HUG), Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jastrow N, Picchiottino P, Savoldelli G, Irion O. [Simulation in obstetrics]. Rev Med Suisse. 2013 Oct 23;9(403):1938-40, 1942. French. PMID 24245015
- [Background] Fransen AF, van de Ven J, Merien AE, de Wit-Zuurendonk LD, Houterman S, Mol BW, Oei SG. Effect of obstetric team training on team performance and medical technical skills: a randomised controlled trial. BJOG. 2012 Oct;119(11):1387-93. doi: 10.1111/j.1471-0528.2012.03436.x. Epub 2012 Aug 13. PMID 22882714
- [Background] Draycott T, Sibanda T, Owen L, Akande V, Winter C, Reading S, Whitelaw A. Does training in obstetric emergencies improve neonatal outcome? BJOG. 2006 Feb;113(2):177-82. doi: 10.1111/j.1471-0528.2006.00800.x. PMID 16411995
- [Background] Crofts JF, Bartlett C, Ellis D, Hunt LP, Fox R, Draycott TJ. Training for shoulder dystocia: a trial of simulation using low-fidelity and high-fidelity mannequins. Obstet Gynecol. 2006 Dec;108(6):1477-85. doi: 10.1097/01.AOG.0000246801.45977.c8. PMID 17138783
- [Background] Deering S, Poggi S, Macedonia C, Gherman R, Satin AJ. Improving resident competency in the management of shoulder dystocia with simulation training. Obstet Gynecol. 2004 Jun;103(6):1224-8. doi: 10.1097/01.AOG.0000126816.98387.1c. PMID 15172856
- [Background] Hickok DE, Gordon DC, Milberg JA, Williams MA, Daling JR. The frequency of breech presentation by gestational age at birth: a large population-based study. Am J Obstet Gynecol. 1992 Mar;166(3):851-2. doi: 10.1016/0002-9378(92)91347-d. PMID 1550152
- [Background] Hannah ME, Hannah WJ, Hewson SA, Hodnett ED, Saigal S, Willan AR. Planned caesarean section versus planned vaginal birth for breech presentation at term: a randomised multicentre trial. Term Breech Trial Collaborative Group. Lancet. 2000 Oct 21;356(9239):1375-83. doi: 10.1016/s0140-6736(00)02840-3. PMID 11052579
- [Background] Collaris RJ, Oei SG. External cephalic version: a safe procedure? A systematic review of version-related risks. Acta Obstet Gynecol Scand. 2004 Jun;83(6):511-8. doi: 10.1111/j.0001-6349.2004.00347.x. PMID 15144330
- [Background] Bogner G, Xu F, Simbrunner C, Bacherer A, Reisenberger K. Single-institute experience, management, success rate, and outcome after external cephalic version at term. Int J Gynaecol Obstet. 2012 Feb;116(2):134-7. doi: 10.1016/j.ijgo.2011.09.027. Epub 2011 Dec 9. PMID 22169098
- [Background] Teoh TG. Effect of learning curve on the outcome of external cephalic version. Singapore Med J. 1997 Aug;38(8):323-5. PMID 9364883
- [Background] Pichon M, Guittier MJ, Irion O, Boulvain M. [External cephalic version in case of persisting breech presentation at term: motivations and women's experience of the intervention]. Gynecol Obstet Fertil. 2013 Jul-Aug;41(7-8):427-32. doi: 10.1016/j.gyobfe.2012.09.029. Epub 2012 Oct 25. French. PMID 23102577